CLINICAL TRIAL: NCT07309328
Title: Evaluation of the Effectiveness of a Cardiac Coherence Exercise on MRI Success and Image Quality in Claustrophobic Patients
Acronym: COCARI
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MLC_2025_6
Record Dates: First submitted 2025-12-04; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Claustrophobia; MRI
MeSH Terms: conditions — Claustrophobia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac Coherence Breathing Exercise During MRI (Experimental): Participants in this arm will undergo their MRI scan while a guided cardiac coherence breathing exercise is played via audiovisual support (screen and headphones) throughout the procedure.
  Interventions: Behavioral: cardiac coherence
- Standard Care During MRI (No Intervention): Participants in this arm will receive standard care during their MRI scan. As per routine clinical practice, children will be offered to watch a cartoon, and adults will be offered to listen to music during the examination. No specific breathing or relaxation exercise will be provided.

INTERVENTIONS:
Behavioral: cardiac coherence — The exercise consists of slow, rhythmic breathing guided by visual and auditory cues designed to induce a state of physiological calm.
  Arms: Cardiac Coherence Breathing Exercise During MRI

SUMMARY:
Claustrophobia, an intense fear of confined spaces, can significantly impair the success of MRI examinations by causing patient movement or early termination of the scan, leading to poor image quality. Cardiac coherence, a breathing technique aimed at synchronizing heart rate and reducing anxiety, has shown benefits in stress management. This randomized controlled trial aims to evaluate whether the use of a guided cardiac coherence exercise during MRI can improve exam success rates and image quality in self-reported claustrophobic patients compared to standard care (cartoons for children, music for adults). The primary outcome is the proportion of interpretable MRI scans with good-quality images, assessed blindly by a radiologist. Secondary outcomes include exam duration, use of the emergency call button, patient satisfaction, and perceived comfort. A total of 220 patients aged 7 years and older will be enrolled over 12 months at the Fondation Adolphe de Rothschild Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 7 years or older
* Undergoing a 1.5T or 3T MRI scan as part of routine care
* Self-reported claustrophobia on the imaging department admission form
* Explicit consent to participate in the study, provided by the patient or a legal representative (for minors)
* Affiliated with or beneficiary of a social security system

Exclusion Criteria:

* Patient under legal protection or guardianship
* Pregnant or breastfeeding woman
* Inability to complete questionnaires and/or perform the cardiac coherence exercise as judged by the investigator

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of interpretable MRI exams with good image quality, rated blindly by a radiologist | Day 1
  This outcome measures the proportion of MRI exams considered interpretable and of good quality, based on image assessment by a radiologist blinded to the intervention group. Any exam for which all planned sequences could not be acquired is considered a failure. Each image is scored on a 5-point scale:
  No artifacts;
  Minor artifacts (edges only), not interfering with interpretation;
  Moderate artifacts, not interfering with interpretation;
  Significant artifacts, partial interpretation possible;
  Major artifacts, hindering interpretation. An exam is considered of good quality if all images are rated as 1 or 2.

IPD SHARING:
Plan to Share IPD: Undecided